CLINICAL TRIAL: NCT04391569
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of Intravenous Ganaxolone in Status Epilepticus
Brief Title: Randomized Therapy In Status Epilepticus
Acronym: RAISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1042-SE-3003
Record Dates: First submitted 2020-04-30; First posted 2020-05-18 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Status Epilepticus
Keywords: Seizure; Status Epilepticus; Convulsive Status Epilepticus; Non-Convulsive Status Epilepticus; Epilepsy
MeSH Terms: conditions — Status Epilepticus; Seizures; Epilepsy | interventions — ganaxolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV Placebo (Placebo Comparator): Placebo bolus dose followed by continuous infusion for 36 hours, followed by 12 hour taper
  Interventions: Drug: Placebo
- IV ganaxolone active (Experimental): Ganaxolone bolus dose followed by continuous infusion for 36 hours, followed by 12 hour taper
  Interventions: Drug: Ganaxolone

INTERVENTIONS:
Drug: Ganaxolone — Ganaxolone will be administered.
  Arms: IV ganaxolone active
Drug: Placebo — Placebo will be administered.
  Arms: IV Placebo

SUMMARY:
This study evaluated the effectiveness and safety of an investigational product (IP), intravenous (IV) ganaxolone, to treat participants with status epilepticus (SE).

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled study to evaluate the efficacy and safety of IV ganaxolone in status epilepticus. Investigational product was added to standard of care following failure of any two or more antiseizure medications (benzodiazepine and one IV antiepileptic drug (AED) or two IV AEDs. Participants were screened for inclusion/exclusion criteria prior to receiving investigational product by continuous IV infusion. Participants were followed for approximately 4 weeks. Participants who are known to be at risk for SE were consented or assented prior to an SE event.

ELIGIBILITY:
Inclusion Criteria:

1. Participant, participant's parent, guardian, or legal authorized representative (LAR) must provide signed of informed consent/assent, and once capable (per institution guidelines), there must be documentation of consent/assent by the participant demonstrating they are willing and aware of the investigational nature of the study and related procedures. Where allowed by law, where the participant lacks the capacity to make informed decisions regarding his/her medical treatment options, the treating clinician may follow their deferred consenting practices. The clinician will make the final decision based on the best interests of the particiapant.
2. Male or females 12 years of age and older at the time of the first dose of IP
3. SE meeting the following criteria:

   a. A diagnosis of SE with or without prominent motor features based on clinical and EEG findings:

   i. Diagnosis is established by:
   * For SE with prominent motor features: Clinical and EEG seizure activity indicative of convulsive, myoclonic or focal motor SE.
   * For SE without prominent motor features (nonconvulsive SE): Appropriate clinical features and an EEG indicative of non-convulsive status epilepticus (NCSE)

   ii. For any type of SE:
   * At least 6 minutes of cumulative seizure activity over a 30-minute period within the hour before IP initiation, AND
   * Seizure activity during the 30 minutes immediately prior to IP initiation

     b. The treating clinician(s) anticipate that IV anesthesia is likely to be the next treatment for SE that persists following initiation of IP
4. Participants must have received any two or more of the following agents for treatment of the current episode of SE administered at an adequate dose and for a sufficient duration, in the judgment of the investigator, to demonstrate efficacy

   * Benzodiazepines,
   * IV Fosphenytoin/phenytoin,
   * IV Valproic acid,
   * IV Levetiracetam,
   * IV Lacosamide,
   * IV Brivaracetam, or
   * IV Phenobarbital
5. Body mass index (BMI) < 40 or, if BMI is not able to be calculated at screening, participant is assessed by investigator as not morbidly obese

Exclusion Criteria:

1. Life expectancy of less than 24 hours
2. Anoxic brain injury or an uncorrected rapidly reversable metabolic condition as the primary cause of SE (e.g., hypoglycemia < 50 milligram per deciliter [mg/dL] or hyperglycemia > 400 mg/dL)
3. Participants who have received high-dose IV anesthetics (e.g., midazolam, propofol, thiopental, or pentobarbital) during the current episode of SE for more than 18 hours, or who continue to have clinical or electrographic evidence of persistent seizures while receiving high-dose IV anesthetics.
4. Clinical condition or advance directive that would NOT permit use of IV anesthesia
5. Participants known or suspected to be pregnant
6. Participants with known allergy or sensitivity to progesterone or allopregnanolone medications/supplements
7. Receiving a concomitant IV product containing Captisol®
8. Known or suspected hepatic insufficiency or hepatic failure leading to impaired synthetic liver function.
9. Known or suspected stage 3B (moderate to severe; estimated glomerular filtration rate [eGFR] 44-30 milliliter/minutes/1.73-meter square [mL/min/1.73m^2]), stage 4 (severe; eGFR 29-15 mL/min/1.73m^2), or stage 5 (kidney failure; eGFR < 15 mL/min/1.73m^2 or dialysis) kidney disease
10. Use of an investigational product for which less than 30 days or 5 half-lives have elapsed from the final product administration. Participation in a non-interventional clinical study does not exclude eligibility.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- United States (53):
  - Marinus Research Site, Birmingham, Alabama
  - Marinus Research Site, Phoenix, Arizona
  - Marinus Research Site, Little Rock, Arkansas
  - Marinus Research Site, Downey, California
  - Marinus Research Site, La Jolla, California
  - Marinus Research Site, Orange, California
  - Marinus Research Site, Sacramento, California
  - Marinus Research Site, Aurora, Colorado
  - Marinus Research Site, Denver, Colorado
  - Marinus Research Site, New Haven, Connecticut
  - Marinus Research Site, Gainesville, Florida
  - Marinus Research Site #1, Miami, Florida
  - Marinus Research Site, Miami, Florida
  - Marinus Research Site, Port Saint Lucie, Florida
  - Marinus Research Site, Tampa, Florida
  - Marinus Research Site, Chicago, Illinois
  - Marinus Research Site, Urbana, Illinois
  - Marinus Research Site, Louisville, Kentucky
  - Marinus Research Site, New Orleans, Louisiana
  - Marinus Research Site, Shreveport, Louisiana
  - Marinus Research Site #1, Baltimore, Maryland
  - Marinus Research Site, Baltimore, Maryland
  - Marinus Research Site, Boston, Massachusetts
  - Marinus Research Site, Worcester, Massachusetts
  - Marinus Research Site, Ann Arbor, Michigan
  - Marinus Research Site, Grand Rapids, Michigan
  - Marinus Research Site, Columbia, Missouri
  - Marinus Research Site, St Louis, Missouri
  - Marinus Research Site, New Brunswick, New Jersey
  - Marinus Research Site, Albuquerque, New Mexico
  - Marinus Research Site, Albany, New York
  - Marinus Research Site, Brooklyn, New York
  - Marinus Research Site, New York, New York
  - Marinus Research Site, Rochester, New York
  - Marinus Research Site, Chapel Hill, North Carolina
  - Marinus Research Site, Charlotte, North Carolina
  - Marinus Research Site, Durham, North Carolina
  - Marinus Research Site, Cincinnati, Ohio
  - Marinus Research Site, Cleveland, Ohio
  - Marinus Research Site, Columbus, Ohio
  - Marinus Research Site, Portland, Oregon
  - Marinus Research Site #1, Philadelphia, Pennsylvania
  - Marinus Research Site #2, Philadelphia, Pennsylvania
  - Marinus Research Site, Philadelphia, Pennsylvania
  - Marinus Research Site, Pittsburgh, Pennsylvania
  - Marinus Research Site, Knoxville, Tennessee
  - Marinus Research Site, Memphis, Tennessee
  - Marinus Research Site, Dallas, Texas
  - Marinus Research Site, Fort Worth, Texas
  - Marinus Research Site, San Antonio, Texas
  - Marinus Research Site, Murray, Utah
  - Marinus Research Site, Richmond, Virginia
  - Marinus Research Site, Madison, Wisconsin
- Australia (4):
  - Marinus Research Site, Randwick, New South Wales
  - Marinus Research Site, South Brisbane, Queensland
  - Marinus Research Site, Box Hill, Victoria
  - Marinus Research Site, Melbourne, Victoria
- Canada (4):
  - Marinus Research Site, Calgary, Alberta
  - Marinus Research Site, Kingston, Ontario
  - Marinus Research Site, Québec, Quebec
  - Marinus Research Site, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a double-blind, randomized, placebo-controlled study that evaluated the efficacy and safety of ganaxolone intravenous (IV) solution in status epilepticus (SE).
Pre-assignment Details: A total of 100 participants were enrolled in the study.
Groups:
- Ganaxolone: Ganaxolone IV administered with a 30-milligrams (mg) bolus dose with initiation of a 36-hour continuous infusion followed by a 12-hour taper.
- Placebo: Placebo IV administered with a bolus and infusion equivalent to volume of IV ganaxolone.
Period: Overall Study
Arm/Group | Ganaxolone | Placebo
Started | 51 | 49
Completed | 30 | 35
Not Completed | 21 | 14
Not completed — Death | 15 | 10
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 3 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Participant discharged to hospice facility | 0 | 1
Not completed — Participant family decision | 1 | 0
Not completed — Participant discharged prematurely | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population comprises all participants who received the investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ganaxolone | Placebo | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (19.40) | 57.0 (19.03) | 57.5 (19.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 30 | 30 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 43 | 43 | 86
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 14 | 27
  White | 34 | 32 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With SE Cessation Within 30 Minutes of Investigational Product (IP) Initiation Without Medications for the Acute Treatment of SE
Description: SE cessation was determined by the investigator based on clinical and electroencephalography (EEG). Medications for the acute treatment of SE were defined as antiepileptic drugs (AEDs) administered to abort ongoing SE or prevent imminent recurrence of SE based on clinical or EEG evidence.
Time Frame: Up to 30 minutes
Population: Intent-To-Treat (ITT) population comprised of all randomized participants in the double-blind phase of the study who received IP and had at least one non-missing efficacy assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 49 | 47
Percentage of participants | 79.59 [65.657 to 89.755] | 12.77 [4.832 to 25.741]
Statistical Analysis 1: Comparison: Ganaxolone vs Placebo; Test type: Other; p = 0.0000, fixed weight combination test — P-value from logistic regression is used for interim data, and Boschloo's test p-value is used for post interim data; P-value is derived by fixed weight (2/3 for interim and 1/3 for post interim) combination test

2. Primary Outcome: Percentage of Participants With no Progression to Intravenous (IV) Anesthesia for 36 Hours Following Investigational Product (IP) Initiation
Description: Percentage of participants with no progression to IV anesthesia for 36 hours following IP initiation SE cessation was based on investigator report with confirmation by assessment of concomitant medication data.
Time Frame: Up to 36 hours after IP initiation
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 49 | 47
Percentage of participants | 63.27 [48.288 to 76.578] | 51.06 [36.064 to 65.924]
Statistical Analysis 1: Comparison: Ganaxolone vs Placebo; Test type: Other; p = 0.1619, fixed weight combination test — P-value from logistics regression is used for interim data, and Boschloo's test p-value is used for post interim data; P-value is derive by fixed weight (2/3 for interim and 1/3 for post interim) combination test

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant who has been administered a pharmaceutical product; it does not necessarily have a causal relationship with this treatment. Treatment-emergent adverse event (TEAE) is defined as an AE that occurred or worsened at the time of or following IP initiation.
Time Frame: Up to 4 weeks after IP initiation
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 51 | 49
Participants
  Any TEAE | 48 | 43
  Serious TEAEs | 19 | 18
  TEAE Leading to study drug discontinuation | 1 | 2
  TEAE leading to withdrawal | 2 | 0
  TEAE resulting in death | 11 | 11

4. Secondary Outcome: Percentage of Participants With no Progression to IV Anesthesia for 72 Hours Following IP Initiation
Description: Percentage of participants with no progression to IV anesthesia for 72 hours following IP initiation SE cessation was assessed by the investigator based on clinical and EEG features.
Time Frame: Up to 72 hours after IP initiation
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 49 | 47
Percentage of participants | 51.02 [36.338 to 65.575] | 46.81 [32.112 to 61.922]
Statistical Analysis 1: Comparison: Ganaxolone vs Placebo; Test type: Other; p = 0.2097, fixed weight combination test

5. Secondary Outcome: Time to SE Cessation Following IP Initiation
Description: Time to SE cessation was assessed for the first 72 hours following IP using the Kaplan-Meier method.
Time Frame: Up to 72 hours after IP initiation
Population: ITT population
Measure: Median (Full Range); unit: hours
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 49 | 47
hours | 0.07 [0.0 to 5.4] | 2.85 [0.0 to 40.8]
Statistical Analysis 1: Comparison: Ganaxolone vs Placebo; Test type: Other; p = 0.0000, Log Rank

6. Secondary Outcome: Percentage of Participants With Any Escalation of Treatment in the First 24 Hours Following IP Initiation
Description: SE cessation will be determined by the investigator based on clinical and EEG. Percentage of participants with any escalation of treatment in the first 24 hours following IP initiation, i.e. any medication other than IP administered for the acute treatment of SE in the first 24 hours following IP initiation was summarized
Time Frame: Up to 24 hours after IP initiation
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 49 | 47
Percentage of participants | 55.10 [40.231 to 69.335] | 80.85 [66.740 to 90.851]
Statistical Analysis 1: Comparison: Ganaxolone vs Placebo; Test type: Other; p = 0.0075, fixed weight combination test — P-value is derived by fixed weight (2/3 for interim and 1/3 for post interim) combination test. P-value from logistics regression is used for interim data, and Boschloo's test p-value is used for post interim data

7. Secondary Outcome: Time to Treatment Escalation in the First 24 Hours Following IP Initiation
Description: For time to treatment escalation (any mediation used for acute treatment of SE), the estimates are based descriptive statistics on participants with treatment escalation in the first 24 hours following IP initiation. For participants without treatment escalation, the time to treatment escalation was censored at IP completion, or discontinuation from the study or death, whichever occurs earlier. The median time to treatment escalation has been presented.
Time Frame: Up to 24 hours after IP initiation
Population: ITT population. Participants with treatment escalation following IP initiation were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 27 | 37
hours | 5.42 [0.5 to 21.6] | 2.32 [0.3 to 20.1]

8. Secondary Outcome: Time to Initiation of Anesthesia for SE Treatment Through the Final Study Follow-up Visit/Contact
Description: Time to initiation of anesthesia for SE treatment through the final study follow-up visit/contact, were calculated based on descriptive statistics. The estimate was censored at study discontinuation, death, or last follow-up of the participant, whichever occurs first. The median time to initiation of anesthesia has been presented.
Time Frame: Up to 4 Weeks following IP initiation
Population: ITT population. Participants who initiated anesthesia for SE treatment were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 22 | 25
hours | 15.00 [1.5 to 417.2] | 3.17 [0.6 to 202.7]

9. Secondary Outcome: Percentage of Participants Who Develop Super Refractory Status Epilepticus (SRSE) Through the Final Study Follow-up Visit/Contact
Description: Percentage of participants who developed SRSE through the final study follow-up visit/contact was provided for each treatment group.
Time Frame: Up to 4 Weeks following IP initiation
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 49 | 47
Percentage of participants | 22.45 [11.774 to 36.624] | 25.53 [13.945 to 40.350]

10. Secondary Outcome: Percent Change From Baseline in Seizure Burden Through 72 Hours Following IP Initiation
Description: The seizure burden through 72 hours following IP initiation is described as the percent of time during which there is electrographic seizure activity from IP initiation to 72 hours. The change from baseline of seizure burden was summarized using descriptive statistics by treatment group. The baseline seizure burden is defined for 30 minutes prior to IP initiation.
Time Frame: Up to 72 hours after IP initiation
Population: ITT population. Participants with percent change from Baseline in seizure burden through 72 hours has been presented.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 39 | 30
Percent change | -59.1 (88.98) | -93.9 (19.79)

ADVERSE EVENTS:
Time Frame: Up to 4 Weeks
Description: Serious adverse events and non-serious adverse events were collected in Safety Population.
Groups:
- Placebo: Participants were randomized 1:1 to receive placebo bolus dose followed by continuous infusion for 36 hours, followed by 12-hour taper
- Ganaxolone: Participants were randomized 1:1 to receive Ganaxolone at various intervals during Day 1 and Day 2.
Arm/Group | Placebo | Ganaxolone
All-Cause Mortality (participants affected / at risk) | 11/49 | 15/51
Serious Adverse Events (participants affected / at risk) | 18/49 | 19/51
Other Adverse Events (participants affected / at risk) | 39/49 | 43/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | Ganaxolone (N=51)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Central nervous system infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (6) | 1 (6)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 1 (1)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Hyperammonaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1) | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 5 (5)
Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | Ganaxolone (N=51)
Urinary tract infection (Infections and infestations) | 4 (4) | 10 (10)
Pneumonia (Infections and infestations) | 0 (0) | 5 (6)
Pneumonia serratia (Infections and infestations) | 3 (3) | 0 (0)
Staphylococcal infection (Infections and infestations) | 3 (3) | 0 (0)
Klebsiella infection (Infections and infestations) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 8 (9) | 12 (13)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Shock (Vascular disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 8 (9) | 4 (4)
Hypothermia (General disorders) | 2 (3) | 5 (5)
Generalised oedema (General disorders) | 1 (1) | 2 (2)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Bradycardia (Cardiac disorders) | 3 (3) | 4 (4)
Tachycardia (Cardiac disorders) | 3 (6) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Transaminases increased (Investigations) | 4 (4) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 2 (2)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT04391569/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT04391569/SAP_001.pdf